CLINICAL TRIAL: NCT05872542
Title: Clinical Effectiveness of Silver Diamine Fluoride on Arresting Caries Lesions in Children
Brief Title: SDF Effectiveness on Arresting Caries in Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Abla A Arafa, MD, Associate Professor, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HAPO-02-K-012-2021-11-844
Record Dates: First submitted 2023-05-01; First posted 2023-05-24 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Dental Caries in Children
Keywords: Silver diamine fluoride; Arrested caries; Deciduous teeth
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Silver Diamine Fluoride (SDF) (Experimental): SDF will be applied once to affected carious teeth surfaces at the end of the first visit. Under proper isolation, only gross debris will be removed and SDF will be applied directly to the carious lesion using micro brush according to the manufacturer's instructions.
  Interventions: Drug: Silver Diamine Fluoride (SDF)
- Glass ionomer restoration (GI) (Active Comparator): GI will be applied to carious lesions following the manufacturer's instructions.
  Interventions: Other: Glass Ionomer Restoration (GI)
- Sodium Fluoride varnish with silver nano-particles (NaF-AgNP) (Active Comparator): NaF-AgNP will be applied once to affected carious teeth surfaces at the end of the first visit. Under proper isolation, only gross debris will be removed and NaF-AgNP will be applied directly to the carious lesion using micro brush according to the manufacturer's instructions.
  Interventions: Other: Sodium fluoride varnish with nano-sliver particles (NaF-AgNP)

INTERVENTIONS:
Drug: Silver Diamine Fluoride (SDF) — Proper isolation of the operating field and removal of gross debris. Minimize contact with the gingiva and mucus membrane. Gentle dryness with compressed air. Dip and dab micro brush on the side of the dapper dish. Apply SDF to the affected surface (one drop/ appointment). Gentle dryness with compressed air for one minute. Remove excess SDF with gauze or cotton pellets. Continue to isolate the site for up to three minutes.
  Arms: Silver Diamine Fluoride (SDF)
Other: Glass Ionomer Restoration (GI) — Application of GI restoration necessitates removal of carious tissue using round bur rotating on low-speed contra and excavation of infected carious dentin. Followed by restoring the prepared cavity with glass ionomer restoration according to the manufacturer's instructions. The restoration will be checked for any high spots and occlusal interference (if any) will be corrected.
  Arms: Glass ionomer restoration (GI)
Other: Sodium fluoride varnish with nano-sliver particles (NaF-AgNP) — Proper isolation of the operating field and removal of gross debris. Minimize contact with the gingiva and mucus membrane. Gentle dryness with compressed air. Dip and dab micro brush on the side of the dapper dish. Apply NaF-AGNP to the affected surface (one drop/ appointment). Gentle dryness with compressed air for one minute. Continue to isolate the site for up to three minutes.
  Arms: Sodium Fluoride varnish with silver nano-particles (NaF-AgNP)

SUMMARY:
Purpose: To assess the clinical effectiveness of silver diamine fluoride (SDF) to control asymptomatic cavitated carious lesions compared to conventional glass ionomer restoration in preschool children.

DETAILED DESCRIPTION:
1. Introduction The global spread of COVID-19 has led to drastic modifications affecting different fields including the field of Pediatric Dentistry. The last emergent guidelines of dental caries management under and following the current pandemic status, specifically recommended minimization of Aerosol Generating Procedures (AGP) and shifting to non- and minimally invasive biological approaches for dental caries management like the use of Silver Diamine Fluoride (SDF).

   In addition, convincing young children to cooperate during conventional restorative dental procedures could be stressful and usually challenging, where the dentist might be compelled to use advanced behavior management techniques such as sedation or general anesthesia.

   The application of SDF focused on arresting and preventing dental caries progression, particularly in children. A high success rate was reported following SDF treatment in arresting dental caries progression. SDF treatment is also considered of low-cost, easy application technique, does not require extensive caries removal, and thus omits the need for local anesthesia administration.

   The SDF clinical effectiveness is obtained through a series of chemical reactions that promote carious lesion arrest. Silver ions possess a bactericidal effect via the inhibition of bacterial cell wall synthesis and DNA synthesis resulting in the disruption of plaque biofilm formation. Both silver and fluoride ions in SDF synergistically enhance remineralization of affected tooth structure and formation of fluorapatite, silver phosphate, and calcium fluoride compounds; hence termed "Silver-fluoride pullet" to arrest dental caries. The formed precipitate not only causes occlusion of the dentinal tubules but also reduces collagen degradation following caries affection. Furthermore, the sustained bactericidal effect of SDF arises from the ability of silver-affected bacteria to kill living bacteria of the same species as they come into contact which is known as the "Zombie phenomenon".

   However, SDF treatment has the side effect of staining everted carious lesions permanently black as a result of the precipitation of silver protein and silver phosphate complexes which could represent a barrier to its application. However, most parents compromise esthetics when their children are subjected to an invasive approach to dental caries management particularly under general anesthesia.

   The use of conventional glass ionomer dental restorations has been frequently used to restore known to have a potent ability to release fluoride which aids in enhancing the remineralization of dental caries and further reduction in the development of new carious lesions. In addition, it is provided in various shades making it a more esthetically appealing dental restoration. However, its application technique necessitates a degree of compliance that could be challenging in young children.

   Thereby, this study will focus on the assessment of the clinical effectiveness of SDF treatment on cavitated carious lesions in preschool children compared to conventional glass ionomer restoration.
2. Materials and methods

2.1. Study design This clinical study will be conducted on a convenient sample of pre-school children attending the Pediatric Dental Clinics, at the College of Dentistry, Umm AlQura University, seeking oral and dental care. Children and their guardians will receive a comprehensive explanation of the dental procedure and expected complications, in addition to the declaration of possible treatment alternatives. A voluntary approval of written consent is required for child participation in this study.

2.2. Sample size calculation The estimation of the sample size relays on that SDF treatment can arrest caries at a rate of 80 percent, with a 10 percent difference to reach clinical significance, at statistical power of 80 percent and the statistical significance level equals 5 percent (α =0.05). Using ClinCalc.com (https://clincalc.com/Stats/SampleSize.aspx), the results showed that 199 carious surfaces per test group will be required. Considering the 10 percent dropout rate at the reassessment time, a minimum of 220 carious teeth surfaces per group will be needed for this study. The average caries tooth surface in children is estimated to be about four surfaces, thus, 60 participants per group will be included in this study.

2.3. Participants' grouping Participants will be randomly assigned using closed envelops distributed by the clinic receptionist, into one of the following groups; Group A: who will receive SDF treatment at the baseline and at Week 24. Group B: who will receive conventional glass ionomer restoration following manufacturer instructions.

2.4. Study procedures Parents will be asked to complete a questionnaire to assess family sociodemographic characteristics. The participants will receive a simple explanation regarding the dental application of SDF, indications, merits, demerits, and barriers to conventional restorative dental treatment as a child crying, screaming, or kicking. Standard sets of high-quality colored pictures that displayed cases of primary and permanent teeth, before and after treatment using SDF for comparison, will be shown to the participants and their parents.

All participants will receive a thorough clinical examination using a disposable dental mirror and ball-end community periodontal index probe. The following will be assessed at the first visit (base record) and at the end of six months (follow-up record):

1. Dental caries experience: using dmfs index (decayed, missing due to caries and filled deciduous tooth surfaces) and the caries lesion extent (ICDAS codes from 3- to 5).
2. Caries activity: arrested or active.
3. Caries risk susceptibility using CariScreen meter.
4. Plaque and gingival indexes will also be scored to assess oral hygiene status.
5. Stimulated saliva will be collected to estimate salivary flow rate and saliva pH.

At the end of the first visit, each participant will receive strict instructions toward guided oral hygiene practice using a dental model.

2.5. Statistical analysis Continuous variables will be summarized with means and standard deviations, and categorical variables will be summarized with counts and percentages.

All data will be analyzed using the SPSS (version 16.0) software package (SPSS Inc., Chicago IL, USA). The significance level will be tested at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children without a history of serious systemic conditions necessitating chronic use of medications.

  * Children whose dental examination reveals at least one untreated asymptomatic cavitated carious lesion (ICDAS index: code 3-5) affecting primary molars.
  * Absence of former history of spontaneous pain from the offending tooth/teeth.
  * Teeth with normal vital pulp response when assessed using sensibility test and absence of any signs of irreversible pulpitis or necrotic pulp degeneration.
  * Absence of abnormal grade of tooth mobility, swelling, or tenderness on palpation or percussion.
  * Absence of any evidence of peri-radicular pathosis, or internal- or external resorption on radiographic examination.

Exclusion Criteria:

* Patients with proven allergy to silver compounds or any component of dental materials to be applied.
* Patients or guardians who refuse to participate in the study or had poor acceptance of SDF treatment.
* Patients with ulcerative gingivitis or stomatitis.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Dental Caries Lesions using ICDAS score at Week 24 | Baseline and Week 24
  The International Caries Detection and Assessment System (ICDAS) is a validated instrument that measures the surface changes of carious lesions by relying on surface characteristics. The ICDAS detection codes for coronal caries range from 0 to 6 depending on the severity of the lesion; code 0: sound tooth surface, code 1:white brown opacity affecting pit or fissure, code 2:distinct changes detected in wet-enamel, code 3: localized enamel breakdown, code 4: underlying dark shadow from dentine, code 5: distinct cavity in dentine, code 6: distinct cavity (more than half surface) in dentine.
Mean Change from Baseline in Dental Caries Lesions using dmfs index at Week 24 | Baseline and Week 24
  The dmfs index is a validated tool that is used to assess the extent of dental caries experience affecting deciduous dentition where "d" stands for decayed, "m" stands for missing tooth due to caries, and "f" stands for filled tooth due to caries.
Change from Baseline in Dental Caries Activity using Arrested or Active caries characteristics at Week 24 | Baseline and Week 24
  Changing of affected carious lesion texture and color; from soft, rough yellow or brown lesion(active caries), to hard smooth dark brown to black color(arrested caries).
Mean Change from Baseline in Dental Caries Susceptibility using the CariScreen Caries Susceptibility Testing meter at Week 24 | Baseline and Week 24
  CariScreen meter is a validated tool that measures adenosine triphosphate-driven bioluminescence for quantification of plaque bacteria to determine if the participant is at low risk (from 0- to 1500 RLUs) or at risk (from1501- to 9999 RLUs) of developing dental caries.

SECONDARY OUTCOMES:
Mean Change from Baseline in oral health status using the Plaque index score at Week 24. | Baseline and Week 24
  The Plaque index is a validated tool to assess plaque accumulation on a scale from 0- to 3, where score 0 indicates the absence of plaque while score 3 denotes plaque deposits covering more than half of the tooth clinical crown
Mean Change from Baseline in oral health status using the Gingival index score at Week 24. | Baseline and Week 24
  The Gingival index is a validated tool to assess the gingival condition on a scale from 0- to 3, as follows: no gingival inflammation (<0.1), mild inflammation (0.1-1.0), moderate inflammation (1.1-1.9), and severe inflammation in case of marked gingival redness and edema with spontaneous bleeding and ulceration (2.0-3.0).
Mean Change from Baseline in saliva pH using pH meter at Week 24. | Baseline and Week 24
  The pH meter is a validated tool to assess the pH of saliva. Stimulated saliva will be collected over five minutes and the saliva pH will be assessed immediately after collecting the saliva sample.

CONTACTS AND LOCATIONS:
Overall Officials: Abla Arafa, Principal Investigator — Assistant Professor
Locations (1):
- UmmAlQuraUniversity, Mecca, Saudi Arabia

REFERENCES:
- [Background] Al-Halabi M, Salami A, Alnuaimi E, Kowash M, Hussein I. Assessment of paediatric dental guidelines and caries management alternatives in the post COVID-19 period. A critical review and clinical recommendations. Eur Arch Paediatr Dent. 2020 Oct;21(5):543-556. doi: 10.1007/s40368-020-00547-5. Epub 2020 Jun 16. PMID 32557183
- [Background] Brian Z, Weintraub JA. Oral Health and COVID-19: Increasing the Need for Prevention and Access. Prev Chronic Dis. 2020 Aug 13;17:E82. doi: 10.5888/pcd17.200266. PMID 32790606
- [Background] BaniHani A, Gardener C, Raggio DP, Santamaria RM, Albadri S. Could COVID-19 change the way we manage caries in primary teeth? Current implications on Paediatric Dentistry. Int J Paediatr Dent. 2020 Sep;30(5):523-525. doi: 10.1111/ipd.12690. No abstract available. PMID 32722881
- [Background] Blumer S, Costa L, Peretz B. Success of Dental Treatments under Behavior Management, Sedation and General Anesthesia. J Clin Pediatr Dent. 2017;41(4):308-311. doi: 10.17796/1053-4628-41.4.308. PMID 28650778
- [Background] Mabangkhru S, Duangthip D, Chu CH, Phonghanyudh A, Jirarattanasopha V. A randomized clinical trial to arrest dentin caries in young children using silver diamine fluoride. J Dent. 2020 Aug;99:103375. doi: 10.1016/j.jdent.2020.103375. Epub 2020 May 16. PMID 32428523
- [Background] Raskin SE, Tranby EP, Ludwig S, Okunev I, Frantsve-Hawley J, Boynes S. Survival of silver diamine fluoride among patients treated in community dental clinics: a naturalistic study. BMC Oral Health. 2021 Jan 20;21(1):35. doi: 10.1186/s12903-020-01379-x. PMID 33472613
- [Background] Fung MHT, Duangthip D, Wong MCM, Lo ECM, Chu CH. Randomized Clinical Trial of 12% and 38% Silver Diamine Fluoride Treatment. J Dent Res. 2018 Feb;97(2):171-178. doi: 10.1177/0022034517728496. Epub 2017 Aug 28. PMID 28846469
- [Background] Peng JJ, Botelho MG, Matinlinna JP. Silver compounds used in dentistry for caries management: a review. J Dent. 2012 Jul;40(7):531-41. doi: 10.1016/j.jdent.2012.03.009. Epub 2012 Apr 3. PMID 22484380
- [Background] Mei ML, Ito L, Cao Y, Li QL, Lo EC, Chu CH. Inhibitory effect of silver diamine fluoride on dentine demineralisation and collagen degradation. J Dent. 2013 Sep;41(9):809-17. doi: 10.1016/j.jdent.2013.06.009. Epub 2013 Jun 27. PMID 23810851
- [Background] Rosenblatt A, Stamford TC, Niederman R. Silver diamine fluoride: a caries "silver-fluoride bullet". J Dent Res. 2009 Feb;88(2):116-25. doi: 10.1177/0022034508329406. PMID 19278981
- [Background] Wakshlak RB, Pedahzur R, Avnir D. Antibacterial activity of silver-killed bacteria: the "zombies" effect. Sci Rep. 2015 Apr 23;5:9555. doi: 10.1038/srep09555. PMID 25906433
- [Background] Seifo N, Robertson M, MacLean J, Blain K, Grosse S, Milne R, Seeballuck C, Innes N. The use of silver diamine fluoride (SDF) in dental practice. Br Dent J. 2020 Jan;228(2):75-81. doi: 10.1038/s41415-020-1203-9. PMID 31980777
- [Background] Zhi QH, Lo EC, Lin HC. Randomized clinical trial on effectiveness of silver diamine fluoride and glass ionomer in arresting dentine caries in preschool children. J Dent. 2012 Nov;40(11):962-7. doi: 10.1016/j.jdent.2012.08.002. Epub 2012 Aug 11. PMID 22892463
- [Background] Llodra JC, Rodriguez A, Ferrer B, Menardia V, Ramos T, Morato M. Efficacy of silver diamine fluoride for caries reduction in primary teeth and first permanent molars of schoolchildren: 36-month clinical trial. J Dent Res. 2005 Aug;84(8):721-4. doi: 10.1177/154405910508400807. PMID 16040729
- [Background] Young DA, Novy BB, Zeller GG, Hale R, Hart TC, Truelove EL; American Dental Association Council on Scientific Affairs; American Dental Association Council on Scientific Affairs. The American Dental Association Caries Classification System for clinical practice: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2015 Feb;146(2):79-86. doi: 10.1016/j.adaj.2014.11.018. PMID 25637205
- [Background] Ekstrand KR, Zero DT, Martignon S, Pitts NB. Lesion activity assessment. Monogr Oral Sci. 2009;21:63-90. doi: 10.1159/000224213. Epub 2009 Jun 3. PMID 19494676